CLINICAL TRIAL: NCT03624205
Title: To Evaluate the Long Term Safety and Efficacy of Drug Coated Balloon SeQuent® Please in Chinese Coronary Instent Restenosis Patients,a Prospective, Multi-center,Randomization Clinical Trial.
Brief Title: The Safety and Efficacy of SeQuent® Please in Real World Chinese Coronary Instent Restenosis Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: B. Braun Medical International Trading Company Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: AAG-O-H-1414
Record Dates: First submitted 2018-08-07; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Coronary In Sentrestenosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: paclitaxel-releasing coronary balloon (SeQuent® Please) — SeQuent® Please with a length of 10mm,15mm,17mm,20mm and 26mm and diameter of 2.5 mm, 2.75 mm, 3.0mm, 3.5mm and 4.0mm are to be used in the trial

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of paclitaxel -eluting PTCA- balloon (SeQuent® Please) in real world Chinese Coronary In Sentrestenosis patients

ELIGIBILITY:
Inclusion Criteria:

Criteria related to subjects

* At the age of 18-80, Both male and female;
* Patients with coronary In sentrestenosis and suitable for the theory of Drug Eluting PTCA Balloon Catheter（SeQuent® Please）, no more than 1 target lesion in each coronary artery
* After pre-dilation of target lesion, the residual stenosis is ≥ 30% , patients with type B dissection
* Patients must agree to sign the ICF and to undergo the clinical follow-up at 30 days, 6 months, 6 months, 12 months, 24 months, 36months, 48 months and 60 months after operation Criteria related to lesions
* The target lesion length and target vessel diameter should be consistent with the instructions of Drug Eluting PTCA Balloon Catheter（SeQuent® Please）

Exclusion Criteria:

Criteria related to subjects

* Women with pregnancy or lactation
* Patient with cardiac shock
* Patients with Hemorrhagic physique or active gastrointestinal ulcers, with cerebral apoplexy or transient cerebral ischemia within 3 months, who couldn't be tolerated the expected aspirin and/or clopidogrel theory
* Patients with severe valvular heart disease
* Patients with severe congestive heart failure or NYHA class IV heart failure;
* Patients who have received heart transplant;
* Patients with life expectancy more than 60 months, or those who is difficulties in clinical follow-up.
* Patients who are currently involved in any other clinical trial;
* Patients that the investigators think that those are not suitable Criteria related to lesions
* Chronic total occlusion
* Lesion that cannot be treated with PTCA or other interventional techniques;
* The vessel diameter < 2.25 mm
* Left main disease needed to be treated Exclusion criteria related to concomitant medication
* Patients who are intolerant to aspirin and/or clopidogrel or have a history of neutrophilopenia or thrombocytopenia, or patients with severe hepatic insufficiency and contraindicated for clopidogrel.
* Patients who are known to be intolerant or allergic to heparin, contrast agent, paclitaxel, iopromide, rapamycin, polylactic acid - glycolic acid polymer, stainless steel;

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patient with coronary In sentrestenosis
Sampling Method: Non-Probability Sample
Enrollment: 520 (Actual)
Dates: Start 2015-04-24 (Actual); Primary Completion 2022-01-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Target Lesion Failure in 12 months after operation | 1 year
  To measure Target Lesion Failure in 12 months by using angiography